CLINICAL TRIAL: NCT04872088
Title: Impact Evaluation of Integrated Interventions to Reduce Child Wasting in Mali
Brief Title: Integrated Research on Acute Malnutrition in Mali (IRAM-MALI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: UNICEF (Other); World Vision (Other); AFRICSante (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRAM-MALI
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-02

CONDITIONS: Acute Malnutrition in Childhood; Wasting
MeSH Terms: conditions — Cachexia | interventions — Secondary Prevention

STUDY DESIGN:
Intervention Model Description: Non-blinded cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive preventive (BCC on child health and nutrition) and screening services from existing unsupervised Nutrition Activity Support Groups (NASGs) without additional support from the IRAM project. Children with wasting are eligible to be enrolled in the existing national Community Management of Acute Malnutrition (CMAM) program.
- Intervention (Experimental): The intervention group will receive the integrated package of interventions that will be delivered by the NASGs.
  The NASG platform will be strengthened by the IRAM project by increasing their number proportional to the size of the population of the catchment area they serve and by regular formative supervision by NGO and health center staff.
  The package of interventions includes:
  * Social and Behavioral Change Communication by NASGs during home visits and group sessions
  * Monthly delivery of preventive SQ-LNS to children 6-17 months of age
  * Screening and referral of children 6-59 months of age through the introduction of the MUAC family approach (distribution MUAC tapes to families and offering formative supervision by NASGs to enhance measurement quality)
  * Cooking demonstrations for complementary foods using nutrientdense foods in the community.
  Interventions: Behavioral: Strengthened SBCC; Dietary Supplement: Preventive nutritional supplement; Behavioral: Family MUAC; Behavioral: Active screening by NASGs; Behavioral: Intensified followup of children with wasting referred to and enrolled in CMAM treatment; Behavioral: Relapse prevention; Behavioral: Cooking demonstrations

INTERVENTIONS:
Behavioral: Strengthened SBCC — Social and Behavioral Change Communication related to prenatal, postnatal, IYCF practices as well as on the care of young children at several specific ages, hygiene, and health will be delivered during monthly home visits by pairs of NASG members.
  Arms: Intervention
Dietary Supplement: Preventive nutritional supplement — Monthly delivery by NAGS pairs of a nutritional supplement: SQ-LNS, at a dose of 28 bags of 20g per month per beneficiary child. The nutritional supplement is limited to :
  - [6-17]months old children diagnosed as non-wasted (MUAC>=125mm)
  Arms: Intervention
Behavioral: Family MUAC — MUAC screening of children 6 to 59 months of age by family members will be introduced. This will involve distributing Shakir MUAC tapes to all intervention households and training mothers/guardians, or any other family member expressing an interest, in the screening of wasting with the MUAC criterion.
  The training will be carried out by the members of the NASGs and during each home visit, they will be able to ensure that the MUAC measurement technique is well mastered by the mother (or another member) and correct the technique if necessary. They will also explain the procedure to be followed if the child is diagnosed as wasted by a family.
  Arms: Intervention
Behavioral: Active screening by NASGs — Monthly screening by the NASG members of the children they follow, using the MUAC.
  Referral to the health center of [6-17] months old children screened as malnourished (result of MUAC orange or red), and follow-up on referral to confirm child was enrolled.
  Arms: Intervention
Behavioral: Intensified followup of children with wasting referred to and enrolled in CMAM treatment — NASG members will conduct biweekly follow-up visits in the households of children with wasting referred to and enrolled in CMAM treatment programs to ensure adherence to the outpatient treatment schedule.
  Arms: Intervention
Behavioral: Relapse prevention — NASG members will conduct biweekly home visits to monitor the nutritional status of children aged 9 to 17 months who were discharged from CMAM treatment after recovery. NASGs members will provide additional counseling to prevent relapse and screen these children for wasting to detect possible relapse.
  Arms: Intervention
Behavioral: Cooking demonstrations — NASGs members will also be supported by the IRAM project in the organization of cooking demonstrations with nutrient-rich foods in the community, during which passive screening of children will be carried out.
  Arms: Intervention

SUMMARY:
The IRAM MALI impact evaluation uses a cluster-randomized controlled study design to assess the impact of the package of integrated interventions aimed at reducing the longitudinal prevalence of wasting by reducing the incidence of child wasting, enhancing the recovery/cure rate from wasting treatment and reducing the relapse rate determined three months after post-treatment recovery from wasting. These interventions include, among other things, strengthening of community care groups (NASGs); home visits with delivery of behavioral change communication about nutrition, health and hygiene (WASH) for young children; distribution of a preventive nutritional supplement; and improved coverage of wasting screening (family MUAC and community screening), management, adherence to treatment and prevention of relapse in the health district of Koutiala, Sikasso region, Mali, West Africa.

DETAILED DESCRIPTION:
Progress in reducing the burden of child wasting is hampered by several factors. First, programmatic evidence on how to prevent wasting is limited. There is a growing body of evidence on the effectiveness of dietary supplements in preventing wasting, but little is known about the effectiveness of other strategies such as behavior change communication (BCC) (with or without supplements), cash transfers, or water, hygiene, and sanitation (WASH) interventions. Second, coverage of CMAM (Community based Management of Acute Malnutrition) treatment remains low in many settings. On the supply side, documented constraints include the complexity of current treatment procedures, which disproportionately affects resource-limited settings, and frequent shortages of treatment commodities. On the demand side, low participation in screening and low treatment uptake and adherence are key constraints to effective treatment.

Reducing the burden of wasting effectively requires coordination and integration of sequenced interventions and services along the continuum of care of child wasting including prevention, screening of cases, the timely and adequate treatment of wasted children, and the prevention of relapse of recovered children.

The overall objective of the study is to assess the impact of an integrated package covering the continuum of care of wasting on the longitudinal prevalence of child wasting.

The implementation of these interventions is led by World Vision Mali in collaboration with the health services of the Koutiala health district (Sikasso region, Mali) and UNICEF, and will take place at health center and community level, and includes i) a prevention component combining the strengthening of Nutrition Activity Support Groups (NASG) (who will conduct monthly home visits to deliver behavioral change communication, group counselling sessions and cooking demonstrations) and the distribution of Small-Quantity Lipid-based Nutrient Supplements (SQ-LNS) to children over 6 months of age; ii) a component related to strengthening screening and referral that will involve families (MUAC family approach) and screening by NASGs; iii) a treatment component that includes strengthening the national CMAM protocol currently in vigor in Mali and intensive follow-up of cases under treatment by NASGs to enhance adherence to treatment; and iv) a targetted prevention component through intensified follow-up visits by NASGs and the distribution of SQ-LNS to children who recovered from wasting.

The study, designed as a randomized controlled clustered trial, will allocate 45 health center catchment areas to an intervention (n=22) and comparison group (n=23) and will assess the impact of the integrated package of interventions in three different cohort samples

* the longitudinal prevalence of wasting in children between 6 and 14 months of age (cohort 1; n=1,620)
* the recovery rate of children 6-23 months of age enrolled in wasting, MAM and SAM treatment (cohort 2; census of all children enrolled in treatment programs between May and December 2021)
* the incidence of relapse in children aged 9-17 months discharged from wasting, MAM and SAM treatment after recovery (cohort 3; n=945), determined 3 months post-treatment.

ELIGIBILITY:
Cohort 1 (prevention cohort):

Inclusion criteria are:

* 6-6.9 months of age
* Singleton
* The mother must live in the study area from the time of inclusion.
* The consent of the mother or guardian

Exclusion criteria are :

* Congenital malformations that make anthropometric measurements impossible.
* Mother intends to leave the study area before January 2022.

Cohort 2 (treatment cohort):

Inclusion criteria are :

* The child is enrolled in CMAM treatment program.
* The child is between 6 and 23 months of age at inclusion
* Child lives in one of the 45 health center catchment areas in the study area

Cohort 3 (relapse cohort):

Inclusion criteria are:

* Child has been successfully treated for wasting and MAM and has been discharged from CMAM treatment program for at least three months
* The child is between 9 and 17 months at time of measurement.
* The child is singleton.
* The mother must live in the study area from the time of inclusion.
* The consent of the mother or guardian

Exclusion criteria are :

* Congenital malformations that make anthropometric measurements impossible.
* Mother intends to leave the study area before January 2022.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9797 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
The longitudinal prevalence of wasting in children enrolled at the age of 6 months followed monthly until the end of the study (Cohort 1). | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  This indicator is defined for each child as the number of visits during which nutritional wasting is observed divided by the total number of monthly visits made (by the interviewers).
Recovery rate in children enrolled at [6-23] months of age for up to 3 months of treatment and followed through to discharge (Cohort 2) | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came first
  This indicator is defined as the number children who recovered from wasting, MAM and SAM according to national program criteria (WHZ>-2 and MUAC>=125mm and absence of bilateral edema for two consecutive visits, within 12 weeks of enrollment in the CMAM program) divided by the total number of treatment results recorded.
Prevalence of relapse after discharge from CMAM treatment (cohort 3). | Up to 4 months, at three months after discharge from CMAM treatment
  This indicator is defined as the proportion of children (9-17 months of age) with WLZ-score <-2 or MUAC <125 mm or bilateral edema three months after discharge from a CMAM wasting and moderate wasting treatment program

SECONDARY OUTCOMES:
Longitudinal prevalence of MAM (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the number of months with MAM diagnosis divided by the total number of monthly visits made by the survey teams.
Longitudinal prevalence of SAM (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined by the number of months with SAM diagnosis divided by the total number of monthly visits made.
Incidence of Wasting, MAM and SAM (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the number of new cases of wasting, MAM and SAM diagnosed during the monthly visits made by the survey teams.
Hemoglobin concentration of children (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progressio
  measured by hemocue reader (model 301)
Prevalence of anaemia (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progressio
  defined as the proportion of children with a hemoglobin level below 11g/dl at the end of the study
Child weight (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Child weight measured by survey teams
Child length (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Child length measured by survey teams
Length-for-age Z-score (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Length-for-age Z-score relative to the 2006 WHO reference
Prevalence of child stunting (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Proportion of children with Length-for-age Z-score (LAZ)<-2 (according to the 2006 WHO reference) at the end of the study
Longitudinal wasting screening coverage (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the proportion of children screened (using MUAC, WLZ or bilateral edema) in the month prior to the monthly visit by the interviewers. Two sub-outcomes will also be concerned:
  * Coverage of screening performed by NASGs in the past month.
  * Coverage of the family MUAC component, which is the screening performed by a family member in the past month.
Referral rate of positive screenings (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the proportion of children tested positive during the month (as reported by the mother) who were referred to the health center or Community health worker's site for treatment.
Early Child development (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  assessed via the Development Milestones Checklist-III score at the end of the study.
Linear growth rate (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  * The change in length per month
  * The change in the LAZ per month
Ponderal growth rate (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  * Weight change per month
  * The change in the WLZ per month
MUAC growth rate (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  change in MUAC per month
  * Weight change per month
  * The change in the WLZ index per month
  * MUAC gain (change in MUAC per month)
Longitudinal prevalence of child morbidity (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined by the number of days with symptoms of acute respiratory infections, fever, diarrhea (three or more loose or liquid stools per day) and malaria divided by the total number of days observed/reported in the recall period
Parental knowledge of nutrition, WASH, and health best practices (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  expressed as cumulative total and domain-specific scores
Longitudinal prevalence of Introduction of (semi) solid and soft complementary foods (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  the proportion of children 6-8 months of age who consumed (semi) solid and soft complementary foods the day before the survey
Longitudinal prevalence of minimum dietary diversity of infant and young children (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  The proportion of children who consumed at least 5 of the 8 food groups (including breast milk) the day before the survey.
Longitudinal prevalence of infant and young child minimum meal frequency (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the proportion of children who had eaten the day before the survey: 2 meals for breastfed children 6-8 months, 3 meals for breastfed children 9-23 months, or 4 meals for non-breastfed children 6-23 monthsMinimum meal frequency for children, defined as the proportion of children who had eaten the day before the survey: 2 meals for breastfed children 6-8 months, 3 meals for breastfed children 9-23 months, or 4 meals for non-breastfed children 6-23 months.
  Minimum acceptable diet, defined as the proportion of children with both minimal dietary diversity and minimal meal frequency on the day before the survey.
  Consumption of iron-rich or iron-fortified foods in children.
Longitudinal prevalence of infant and young child minimum acceptable diet (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the proportion of children with both minimal dietary diversity and minimal meal frequency on the day before the survey.
Longitudinal prevalence of continuous breastfeeding (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the proportion of children breastfed during the study
Longitudinal prevalence of infant and young child consumption of iron-rich or iron-fortified foods (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the proportion of children who consumed flesh foods or iron-fortied foods the day before the survey
Vaccination coverage (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Proportion of children with complete vaccination for their age
Adoption of practices recommended by NASGs (cohort 1) | Up to 7 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  related to WASH, treated net use, family planning, deworming, vitamin A, childbirth registration, use of iodized salt, and consumption of SQ-LNS
Weight-for-length Z-score and MUAC at enrollment in CMAM (cohort 2) | Up to 7 months, at the date of inclusion in CMAM program
  weight-for-length Z-score (relative to the 2006 WHO reference) and MUAC(mm)
Duration of CMAM treatment (cohort 2) | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came first
  defined as the number of days spent on treatment (enrollment and discharge) in children 6-23 months of age at enrollment, according to health registers
Treatment adherence (cohort 2) | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came first
  defined as the proportion of cases enrolled for treatment who received timely treatment from dedicated services (health center or Community Health Worker) until recovery
Treatment outcomes (drop-out, death, transfer, non-response rates) (cohort 2) | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came firs
  Among cases of wasting, MAM and SAM enrolledin CMAM treatment
Longitudinal prevalence of childhood morbidity (cohort 2) | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came first
  defined by the number of days with symptoms of acute respiratory infections, fever, diarrhea (three or more loose or liquid stools per day) and malaria divided by the total number of days observed/reported in the recall period
Mid-Upper Arm Circumference of children (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  measured using Shakir MUAC tape by survey teams
Child weight (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  Weight measured by survey teams
Child length(cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  Length measured by survey teams
Weight-for-length Z-score (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  Weight-for-length Z-score relative to the 2006 WHO reference
Length-for-age Z-score (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  Length-for-age Z-score relative to the 2006 WHO reference
Child Stunting (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  defined as the proportion of children with Length-for-age Z-score <-2 (relative to the 2006 WHO reference)
Wasting screening coverage (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  defined as the proportion of children screened (using MUAC, WLZ-score or bilateral edema) in the month prior to the interviewer's visit. Two sub-outcomes will also be concerned:
  * Coverage of screening performed by NASGs in past month.
  * Coverage of the MUAC family component, which is the screening performed by a family member in past month.
Prevalence of readmission (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  Prevalence of children readmitted to CMAM treatment within three months after discharge from CMAM treatment from MAS and MAM treatment programs.
Prevalence of anemia (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  defined as the proportion of children with a hemoglobin level below 11g/dl
Hemoglobin concentration of children (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  measured by hemocue reader (model 301) by survey teams
Longitudinal prevalence of childhood morbidity (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  defined by the number of days with symptoms of acute respiratory infections, fever, diarrhea (three or more loose or liquid stools per day) and malaria divided by the total number of days observed/reported in the recall period
Prevalence of minimum dietary diversity of infant and young children (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  The proportion of children who consumed at least 5 of the 8 food groups (including breast milk) the day before the survey.
Prevalence of infant and young child minimum meal frequency (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  defined as the proportion of children who had eaten the day before the survey: 2 meals for breastfed children 6-8 months, 3 meals for breastfed children 9-23 months, or 4 meals for non-breastfed children 6-23 monthsMinimum meal frequency for children, defined as the proportion of children who had eaten the day before the survey: 2 meals for breastfed children 6-8 months, 3 meals for breastfed children 9-23 months, or 4 meals for non-breastfed children 6-23 months.
  Minimum acceptable diet, defined as the proportion of children with both minimal dietary diversity and minimal meal frequency on the day before the survey.
  Consumption of iron-rich or iron-fortified foods in children.
Prevalence of infant and young child minimum acceptable diet (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  defined as the proportion of children with both minimal dietary diversity and minimal meal frequency on the day before the survey.
Prevalence of infant and young child consumption of iron-rich or iron-fortified foods (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  defined as the proportion of children who consumed flesh foods or iron-fortied foods the day before the survey
Prevalence of continuous breastfeeding (cohort 1) | Up to 4 months, at three months after discharge from CMAM treatment
  defined as the proportion of children breastfed during the study
Adoption of practices recommended by NASGs (cohort 3) | Up to 4 months, at three months after discharge from CMAM treatment
  related to WASH, treated net use, family planning, deworming, vitamin A, childbirth registration, use of iodized salt, and consumption of SQ-LNS

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Huybregts, PHD, Principal Investigator — IFPRI; Elodie Becquey, PHD, Principal Investigator — IFPRI; Jef Leroy, Principal Investigator — IFPRI
Locations (1):
- Koutiala Health District, Sikasso, Mali

IPD SHARING:
Plan to Share IPD: Yes
In accordance with IFPRI's policy on research data management and open access, at the time of publication of scientific articles presenting results, the fully anonymized databases will become a public good and will be made available to the scientific community, government, and partners.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication of scientific articles presenting results, the fully anonymized databases will become a public good and will be made available to the scientific community, government, and partners.

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT04872088/SAP_000.pdf